CLINICAL TRIAL: NCT00708409
Title: Long-Term Follow-up After the Autograft Aortic Valve Procedure (Ross Operation)-the German-Dutch- Ross Registry
Brief Title: Long-Term Follow-up After the Autograft Aortic Valve Procedure (Ross Operation)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Luebeck (Other)
Responsible Party: Hans Hinrich Sievers, University of Schleswig-Holstein, Campus Lübeck, Clinic for cardiac surgery, University of Schleswig-Holstein, Campus Lübeck, Clinic for cardiac surgery
Other Study IDs: Ross-01
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-01

CONDITIONS: Aortic Valve Disease
Keywords: Ross operation; autograft procedure; pulmonary homograft; root replacement technique; subcoronary implantation technique
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transplantation, Autologous; Transplantation, Homologous

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Autograft operations with the subcoronary technique
  Interventions: Procedure: Cardiac valve surgery
- 2: Autograft operations with the root replacement technique
  Interventions: Procedure: Cardiac valve surgery

INTERVENTIONS:
Procedure: Cardiac valve surgery — Different autograft implantation techniques.
  Other Names: Ross operation, autograft, homograft

SUMMARY:
With the current knowledge of aortic valve replacement modalities, no specific recommendations can be given and the decision for a particular prosthesis or procedure is rather arbitrarily. The investigators hypothesize that the autograft procedure according to Ross is superior in terms of hemodynamic (especially regression of left ventricular hypertrophy) and major adverse valve related events even in a long-term course

DETAILED DESCRIPTION:
For patients with aortic valve disease requiring surgical treatment several options are available. In some instances the valve can be repaired, however replacement of the valve is usually necessary. The choice for a particular aortic valve replacement procedure is influenced by several inter-related factors (e.g. prosthesis, procedure itself, patient age, concomitant disease, atrial fibrillation, center's experience, and preference of the referring cardiologist, the attending surgeon and the patient). Often, more than one type of prosthesis seems suitable for the individual patient, whereby the decision for a particular prosthesis is made rather arbitrarily.

With the current knowledge on outcome of patients after aortic valve replacement with different types of prosthesis (pulmonary autograft according to Ross, bioprosthesis, mechanical heart valve), no specific recommendation can be given. This is especially true for the autograft, since no long-term outcome is yet available from clinical practice.

In 2001 the German Ross Registry was established by our working group. Although the Ross procedure was expected to be a lifelong solution for aortic valve disease, it seemed appropriate to make a collaborative effort to establish a multicenter long term follow-up study to examine longitudinal clinical outcomes associated with the procedure, as well as, attempt to resolve and identify the many technical considerations necessary for successful execution of the procedure. With these issues in mind, we have already included about 1400 Ross operated patients from nine participating centers into the registry with up to fourteen years follow-up. The first release of an annual report was presented in February 2004. The main limitation of this Registry is the limited maximal time span of follow-up keeping in mind that the next years of the follow-up are most important for evaluating the Ross procedure because possible degeneration of the aortic valve substitute may occur.

Therefore long-term observation is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the need for aortic valve replacement, aortic valve replacement in the young with the need of valve growth potential, contraindication to oral anticoagulation therapy, female patients with the wish of childbearing,

Exclusion Criteria:

* Extensive coronary artery disease, extensive aortic root calcification, severely impaired left ventricular function, failure to provide informed consent, current participation in another clinical trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2001-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
all cause reoperation rate | one year

SECONDARY OUTCOMES:
valve-related mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Hinrich Sievers, MD, Principal Investigator — University Schleswig-Holstein, Campus Lübeck, Clinic for cardiac surgery
Locations (1):
- University Clinic of Schleswig Holstein, Campus Luebeck, Lübeck, Germany

REFERENCES:
- [Derived] Aboud A, Charitos EI, Fujita B, Stierle U, Reil JC, Voth V, Liebrich M, Andreas M, Holubec T, Bening C, Albert M, Fila P, Ondrasek J, Murin P, Lange R, Reichenspurner H, Franke U, Gorski A, Moritz A, Laufer G, Hemmer W, Sievers HH, Ensminger S. Long-Term Outcomes of Patients Undergoing the Ross Procedure. J Am Coll Cardiol. 2021 Mar 23;77(11):1412-1422. doi: 10.1016/j.jacc.2021.01.034. PMID 33736823
- [Derived] Charitos EI, Takkenberg JJ, Hanke T, Gorski A, Botha C, Franke U, Dodge-Khatami A, Hoerer J, Lange R, Moritz A, Ferrari-Kuehne K, Hetzer R, Huebler M, Bogers AJ, Stierle U, Sievers HH, Hemmer W. Reoperations on the pulmonary autograft and pulmonary homograft after the Ross procedure: An update on the German Dutch Ross Registry. J Thorac Cardiovasc Surg. 2012 Oct;144(4):813-21; discussion 821-3. doi: 10.1016/j.jtcvs.2012.07.005. Epub 2012 Aug 9. PMID 22883549
- [Derived] Charitos EI, Stierle U, Hanke T, Schmidtke C, Sievers HH, Richardt D. Long-term results of 203 young and middle-aged patients with more than 10 years of follow-up after the original subcoronary Ross operation. Ann Thorac Surg. 2012 Feb;93(2):495-502. doi: 10.1016/j.athoracsur.2011.10.017. Epub 2011 Dec 22. PMID 22197618
- [Derived] Sievers HH, Stierle U, Charitos EI, Hanke T, Misfeld M, Matthias Bechtel JF, Gorski A, Franke UF, Graf B, Robinson DR, Bogers AJ, Dodge-Khatami A, Boehm JO, Rein JG, Botha CA, Lange R, Hoerer J, Moritz A, Wahlers T, Breuer M, Ferrari-Kuehne K, Hetzer R, Huebler M, Ziemer G, Takkenberg JJ, Hemmer W; German-Dutch Ross Registry. Major adverse cardiac and cerebrovascular events after the Ross procedure: a report from the German-Dutch Ross Registry. Circulation. 2010 Sep 14;122(11 Suppl):S216-23. doi: 10.1161/CIRCULATIONAHA.109.925800. PMID 20837916
- [Derived] Sievers HH, Stierle U, Charitos EI, Hanke T, Gorski A, Misfeld M, Bechtel M. Fourteen years' experience with 501 subcoronary Ross procedures: surgical details and results. J Thorac Cardiovasc Surg. 2010 Oct;140(4):816-22, 822.e1-5. doi: 10.1016/j.jtcvs.2009.11.042. Epub 2010 Mar 17. PMID 20299029